CLINICAL TRIAL: NCT04079088
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Phase 2 Study to Evaluate the Efficacy and Safety of Oral BIIB061 as Add-On Therapy to Interferon-Beta 1 or Glatiramer Acetate Therapies in Relapsing Multiple Sclerosis
Brief Title: Study to Evaluate Oral BIIB061 Added to Interferon-beta1 (IFN-β1) or Glatiramer Acetate in Relapsing Multiple Sclerosis (RMS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision to discontinue BIIB061 program was based on lack of stronger preclinical effects of BIIB061 on remyelination relative to opicinumab, that showed limited clinical efficacy in phase 2 clinical studies. This was not related to safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231MS201; 2019-001847-28 (EudraCT Number)
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — Interferon-beta; Interferon beta-1a; peginterferon beta-1a; Interferon beta-1b; Glatiramer Acetate; Coat Protein Complex I

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive BIIB061-matched placebo, orally once daily in addition to IFN-β1 injection or glatiramer acetate for up to 72 weeks.
  Interventions: Drug: Placebo; Biological: Interferon-beta1; Drug: Glatiramer acetate
- BIIB061 Dose 1 (Experimental): Participants will receive BIIB061 Dose 1 orally once daily in addition to IFN-β1 injection or glatiramer acetate for up to 72 weeks.
  Interventions: Drug: BIIB061; Biological: Interferon-beta1; Drug: Glatiramer acetate
- BIIB061 Dose 2 (Experimental): Participants will receive BIIB061 Dose 2 orally once daily in addition to IFN-β1 injection or glatiramer acetate for up to 72 weeks.
  Interventions: Drug: BIIB061; Biological: Interferon-beta1; Drug: Glatiramer acetate
- BIIB061 Dose 3 (Experimental): Participants will receive BIIB061 Dose 3 orally once daily in addition to IFN-β1 injection or glatiramer acetate for up to 72 weeks.
  Interventions: Drug: BIIB061; Biological: Interferon-beta1; Drug: Glatiramer acetate

INTERVENTIONS:
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo
Drug: BIIB061 — Administered as specified in the treatment arm.
  Arms: BIIB061 Dose 1; BIIB061 Dose 2; BIIB061 Dose 3
Biological: Interferon-beta1 — Stable dose as prescribed by the physician.
  Other Names: Avonex, Plegridy, Betaferon/Betaseron, Extavia, or Rebif
Drug: Glatiramer acetate — Stable dose as prescribed by the physician.
  Other Names: Copaxone, Glatopa

SUMMARY:
The primary objectives of the study are to evaluate the safety of BIIB061 versus placebo in participants with Relapsing Multiple Sclerosis (RMS), and to evaluate the efficacy of BIIB061 to improve disability outcome versus placebo in participants with RMS.

The secondary objectives of the study are to evaluate the effects of BIIB061 versus placebo on brain magnetic resonance imaging (MRI) markers of remyelination and axon preservation in chronic Multiple Sclerosis lesions and to evaluate the effects of BIIB061 versus placebo on additional measures of improved disability outcome.

DETAILED DESCRIPTION:
BIIB061's unique mechanism of action may provide a pharmacological intervention to overcome the failure of remyelination in all forms of multiple sclerosis by blocking mechanisms that prevent differentiation of oligodendrocytes progenitors.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with relapsing-remitting multiple sclerosis (RRMS) or secondary progressive multiple sclerosis (SPMS)
* Have a Baseline Expanded Disability Status Scale (EDSS) score of 2.0 to 6.0
* Have a MS disease duration of ≤20 years from first MS symptom(s)
* Must have at least one of the following occurring within 12 months prior to

Day 1/Baseline:

(a) ≥1 clinical relapse(s) or objective disability worsening (as per treating neurologist's judgment) (b) ≥1 Gadolinium (Gd)-enhancing T1 lesion(s) on brain or spinal cord Magnetic Resonance Imaging (MRI) (c) ≥1 new T2 lesion(s) on brain or spinal cord MRI (the reference scan used to detect new T2 lesion formation has to be ≤12 months prior to Day 1/Baseline)

* Must have been taking one of the following disease-modifying therapy (DMTs) at a stable dose for at least 12 weeks prior to Day 1/Baseline:

  1. Interferon-beta1 (IFN-β1): Avonex, Plegridy, Betaferon/Betaseron, Extavia, or Rebif
  2. Glatiramer acetate (Copaxone or Glatopa).

     Key Exclusion Criteria:
* A documented history of clinically significant persistent neutralizing antibody against IFN-β1 (applicable only for participants entering the study with IFN-β1 as a background DMT), in the opinion of the Investigator
* Contraindications to MRI, for example, presence of pacemakers or other implanted metal devices (excluding dental braces), an allergy to Gd, renal impairment, or claustrophobia that cannot be medically managed
* History or a positive test result at Screening for human immunodeficiency virus
* Current hepatitis C infection (defined as positive hepatitis C virus [HCV] antibody and detectable HCV Ribonucleic acid (RNA)). Participants with positive HCV antibody and undetectable HCV RNA are eligible to participate in the study (United States [US] Centers for Disease Control and Prevention)
* Current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] or total hepatitis B core antibody [anti-HBc]). Participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive anti-HBc, and positive hepatitis B surface antibody [anti-HBs]) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) are eligible to participate in the study
* History of systemic hypersensitivity reaction to BIIB061
* History of suicidal ideation or an episode of clinically severe depression (as determined by the Investigator) within 12 weeks of screening
* Clinically significant (as determined by the Investigator) 12-lead ECG or laboratory assessment abnormalities
* Any condition affecting study treatment absorption (e.g., gastrectomy)
* Treatment with statins (3-hydroxy-3-methyl-glutaryl coenzyme A reductase inhibitors) or proprotein convertase subtilisin kexin 9 (PCSK9) inhibitors (e.g., alirocumab and evolocumab) within 8 weeks prior to Day 1/Baseline
* Inability or unwillingness to comply with study requirements
* Other unspecified reasons that, in the opinion of the Investigator or Biogen that make the participant unsuitable for enrollment.

Note: Other protocol defined inclusion/ exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2024-09-18 (Estimated); Study Completion 2024-09-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | First dose of study drug to end of the study (Up to Week 84)
  An AE is any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Overall Disability Response Score (ODRS) at Week 48 | Baseline, Week 48
  ODRS is a multicomponent score based on 4 components: Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), 9-Hole Peg Test in the dominant hand (9HPT-D), and 9HPT in the nondominant hand (9HPT-ND). It assesses overall changes in disability over time. The 4 individual scores are added together to get the overall score that ranges from +4 to -4. At each visit, each component is given a score relative to baseline: -1 if threshold is met for worsening, 0 if no changes meet threshold criteria, or +1 if threshold is met for improvement. The thresholds for T25FW and 9HPT are defined by a 15% change from baseline (≥15% decrease from baseline for improvement and ≥15% increase from baseline for worsening). For EDSS, improvement is defined as a ≥1.0-point decrease in EDSS from a baseline score of ≤6.0, and worsening is defined as a ≥1-point increase from a baseline score of ≤5.5 or a ≥0.5-point increase from a baseline score equal to 6.0.

SECONDARY OUTCOMES:
Change from Baseline in Normalized Magnetization Transfer Ratio (nMTR) at Week 48 | Baseline, Week 48
  Remyelination will be measured using magnetization transfer ratio (MTR) in chronic MS lesion detected on brain MRI.
Change from Baseline in Diffusion Tensor Imaging Radial Diffusivity (DTI-RD) at Week 48 | Baseline, Week 48
  Axon and myelin preservation will be measured using DTI-RD in chronic MS lesions detected on brain MRI.
Change from Baseline in Normalized T1 (nT1) Intensity at Week 48 | Baseline, Week 48
  Remyelination and axon preservation will be assessed by nT1 intensity in chronic MS lesions on brain MRI.
Change from Baseline in T1 Hypointense Volume at Week 48 | Baseline, Week 48
  Remyelination and axon preservation will be assessed by T1 hypointense volume in chronic MS lesions on brain MRI.
Percentage of Participants with 12-week Confirmed Improvement in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND | Up to Week 48
  EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist. The T25FW is a quantitative mobility and leg function performance test based on a timed walk over 25 feet. The score for the T25FW is averaged between two completed trials. The 9HPT is a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs.
Percentage of Participants with 12-week Confirmed Worsening in at Least 1 of the Following Assessments: EDSS, T25FW, 9HPT-D, or 9HPT-ND | Up to Week 48
  EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist. The T25FW is a quantitative mobility and leg function performance test based on a timed walk over 25 feet. The score for the T25FW is averaged between two completed trials. The 9HPT is a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs.
ODRS Accounting Only for 12-week Confirmed Events of Worsening and Improvement on Respective Components over the First 48 Weeks of Treatment | 48 weeks
  ODRS is a multicomponent score based on 4 components: EDSS, T25FW, 9HPT-D, and 9HPT-ND. It assesses overall changes in disability over time. The 4 individual scores are added together to get the overall score that ranges from +4 to -4. At each visit, each component is given a score relative to baseline: -1 if threshold is met for worsening, 0 if no changes meet threshold criteria, or +1 if threshold is met for improvement. The thresholds for T25FW and 9HPT are defined by a 15% change from baseline (≥15% decrease from baseline for improvement and ≥15% increase from baseline for worsening). For EDSS, improvement is defined as a ≥1.0-point decrease in EDSS from a baseline score of ≤6.0, and worsening is defined as a ≥1-point increase from a baseline score of ≤5.5 or a ≥0.5-point increase from a baseline score equal to 6.0.
ODRS using 20% Threshold for T25FW over the First 48 Weeks of Treatment | 48 weeks
  ODRS is a multicomponent score based on 4 components: EDSS, T25FW, 9HPT-D, and 9HPT-ND. It assesses overall changes in disability over time. The 4 individual scores are added together to get the overall score that ranges from +4 to -4. At each visit, each component is given a score relative to baseline: -1 if threshold is met for worsening, 0 if no changes meet threshold criteria, or +1 if threshold is met for improvement. The thresholds for T25FW and 9HPT are a 20% and 15% change from baseline respectively. For EDSS, improvement is defined as a ≥1.0-point decrease in EDSS from a baseline score of ≤6.0, and worsening is defined as a ≥1-point increase from a baseline score of ≤5.5 or a ≥0.5-point increase from a baseline score equal to 6.0.
ODRS using 20% Threshold for T25FW, 9HPTD, and 9HPT-ND over the First 48 Weeks of Treatment | 48 weeks
  ODRS is a multicomponent score based on 4 components: EDSS, T25FW, 9HPT-D, and 9HPT-ND. It assesses overall changes in disability over time. The 4 individual scores are added together to get the overall score that ranges from +4 to -4. At each visit, each component is given a score relative to baseline: -1 if threshold is met for worsening, 0 if no changes meet threshold criteria, or +1 if threshold is met for improvement. The thresholds for T25FW and 9HPT are a 20% change from baseline. For EDSS, improvement is defined as a ≥1.0-point decrease in EDSS from a baseline score of ≤6.0, and worsening is defined as a ≥1-point increase from a baseline score of ≤5.5 or a ≥0.5-point increase from a baseline score equal to 6.0.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/